CLINICAL TRIAL: NCT03623399
Title: Does Laparoscopic Entrance and Intraoperative Intraabdominal Gas Pressure Effect Postoperative Pain Score
Brief Title: Laparoscopic Gas Pressure and Postoperative Pain Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seda Yuksel Simsek (Other)
Responsible Party: Sponsor-Investigator, Seda Yuksel Simsek, Gynecology Specialist, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Baskent University
Record Dates: First submitted 2018-08-05; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain; Laparoscopy
Keywords: postoperative pain; Intraabdominal laparoscopic gas pressure
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15 mmhg-15mmhg (No Intervention): Abdominal entrance pressure will be set to 15 mmhg , after laparoscopic visualization of abdomen ; maintenance pressure will be set to 15 mmhg.
- 15 mmhg-12 mmhg (Other): Abdominal entrance pressure will be set to 15 mmhg , after laparoscopic visualization of abdomen ; maintenance pressure will be set to 12 mmhg.
  Low gas pressure laparoscopy
  Interventions: Procedure: low gas pressure laparoscopy
- 12 mmhg-12 mmhg (Other): Abdominal entrance pressure will be set to 12 mmhg , after laparoscopic visualization of abdomen ; maintenance pressure will be set to 12 mmhg.
  Low gas pressure laparoscopy
  Interventions: Procedure: low gas pressure laparoscopy

INTERVENTIONS:
Procedure: low gas pressure laparoscopy — To apply different CO2 entrance and intraoperative pressures
  Arms: 12 mmhg-12 mmhg; 15 mmhg-12 mmhg

SUMMARY:
Aim of the study is to determine the effect of different laparoscopic intraoperative intraabdominal gas (CO2) pressures on the extent of postoperative pain scores.

DETAILED DESCRIPTION:
In this study investigator planned to randomize patients into three groups ; in the first group abdominal entrance pressure will be 15 mmhg and intraoperative pressure will be 15 mmhg too ; in the second group again entrance pressure will be 15 mmhg , intraoperative pressure will be 12 mmhg ; and in the thirth group both entrance and intraoperative pressures will be 12 mmhg. During operation intraoperative mean pressures will be recorded every 15 minutes , also end tidal CO2 pressures will also assesed by the anesthesiologist. Every participant will take , same standard analgesics ; 2 mg/kg contramal and 1 gr i.v. paracetamol at the end of the operation ; except the ones who has allergy to these analgesics. At postoperative 6 th and 24 th hours patients will be asked to execute the visual analogue score (VAS) form to assess the pain . Only patients with benign gynecologic pathologies will be included in to the study and informed consent forms will be taken from all participants.

ELIGIBILITY:
Inclusion Criteria:

* benign gynecologic pathologies which requires laparoscopic surgery

Exclusion Criteria:

* patients who has malign gynecologic pathologies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain scores | Postoperative 6 th hour
  Difference between pain scores of participitants according to differing gas pressures applied.

CONTACTS AND LOCATIONS:
Overall Officials: Husnu Celık, Prof., Study Chair — Baskent University
Locations (1):
- Seda Yuksel Simsek, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
primary outcomes of the study

REFERENCES:
- [Background] Koc M, Ertan T, Tez M, Kocpinar MA, Kilic M, Gocmen E, Aslar AK. Randomized, prospective comparison of postoperative pain in low- versus high-pressure pneumoperitoneum. ANZ J Surg. 2005 Aug;75(8):693-6. doi: 10.1111/j.1445-2197.2005.03496.x. PMID 16076335